CLINICAL TRIAL: NCT06247163
Title: Prospective PET-guided Radiotherapy for Patients With Small Cell Lung Cancer.
Brief Title: PET-guided Radiotherapy for Patients With Small Cell Lung Cancer.
Acronym: PET-ART
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Maja Guberina, PD Dr. med. (MD) Maja Guberina, specialist in radiation oncology, senior consultant, University Hospital, Essen
Other Study IDs: 23-11560-BO
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: PET based Raditherapy boost — An Interim PET CT will be performed. If there is residual vital tumor, a higher radiation dose will be applied.

SUMMARY:
There is a prospective risk-adapted evaluation of the optimal dose of radiotherapy for definitive radiotherapy of locally advanced small cell lung cancer within the corridor recommended as standard therapy according to the current interdisciplinary S3 guideline of the German Cancer Society/Cancer Aid/AWMF

DETAILED DESCRIPTION:
The main objective of this study is to determine whether patients with SCLC who have a metabolically active residual tumor in the fluorodeoxyglucose (FDG) PET/CT scan after two to three cycles of induction chemotherapy have a similarly low local recurrence rate with higher dose. There is a prospective risk-adapted evaluation of the optimal dose of radiotherapy for definitive radiotherapy of locally advanced small cell lung cancer within the corridor recommended as standard therapy according to the current interdisciplinary S3 guideline of the German Cancer Society/Cancer Aid/AWMF. Allocation to PET boost, if confirmed vital tumor rest by PET CT and biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologic confirmation
* Limited disease

Exclusion Criteria:

* Other histology than small cell lung cancer
* Further tumor diagnosis
* ECOG 3 or worse
* Extensive disease
* stage IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed diagnosis of small cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2025-06-22 (Estimated); Study Completion 2029-06-22 (Estimated)

PRIMARY OUTCOMES:
Local recurrence free survival | 2 months to 5 years
  Local recurrence free survival
Distant recurrence free survival | 2 months to 5 years
  Distant recurrence free survival
Overall survival | 2 months to 5 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Essen, Essen, Germany

IPD SHARING:
Plan to Share IPD: No